CLINICAL TRIAL: NCT00294606
Title: Comparison of the Effects of Phenylephrine and Norepinephrine on Cardiac Function During Carotid Cross-Clamping During Carotid Endarterectomy Under General Anesthesia
Brief Title: Comparison of the Effects of Phenylephrine and Norepinephrine on Cardiac Function During Carotid Artery Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: R-05-941
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Last update posted 2006-02-22 (Estimated); Status verified 2006-02

CONDITIONS: Vasopressor Agents; Endarterectomy, Carotid; Echocardiography, Transesophageal
Keywords: vasopressor agents; carotid endarterectomy; cardiac function; transesophageal echocardiography; wall motion abnormalities
MeSH Terms: interventions — Norepinephrine

INTERVENTIONS:
Drug: Comparison of Effects of Phenylephrine and Norepinephrine

SUMMARY:
This will be a prospective, randomized, double-blinded, cross-over clinical trial to compare the effects of phenylephrine or norepinephrine on cardiac function during carotid artery surgery in patients under general anesthesia. The effect of the vasopressor on cardiac function will be measured using electrocardiography, transesophageal echocardiography and cardiac troponin I intraoperatively and postoperatively. We will use a cross-over pattern since both drugs exhibit rapid onset and short duration of action. We hypothesize that there will be less myocardial ischemia associated with the use of norepinephrine when compared with phenylephrine during carotid artery surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective carotid endarterectomy under general anesthesia
* > 18 years old
* Written informed consent

Exclusion Criteria:

* Contraindication to general anesthesia
* Contraindication to transesophageal anesthesia
* esophageal disease
* esophageal stricture
* history of esophageal or gastric bleeding
* esophageal anatomic abnormality
* past esophageal or gastric surgery
* severe dysphagia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2006-02; Study Completion 2006-02

PRIMARY OUTCOMES:
Myocardial ischemia measures by transesophageal echocardiography and ST segment analyses

SECONDARY OUTCOMES:
Myocardial ischemia measures by cardiac troponin I

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary A Craen, MD, FRCPC, Principal Investigator — Associate Professor University of Western Ontario
Locations (1):
- University Hospital, LHSC, London, Ontario, Canada